CLINICAL TRIAL: NCT02242630
Title: Improvement in Function and Pain Due to Subacromial Bursitis in Relationship to Dose of Triamcinolone Acetonide and Methylyprednisolone
Brief Title: Relationship to Dose of Triamcinolone Acetonide and Methylyprednisolone to Improvement in Subacromial Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FKE20140023H
Record Dates: First submitted 2014-09-14; First posted 2014-09-17 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-08

CONDITIONS: Subacromial Bursitis; Shoulder Pain
Keywords: Subacromial bursitis; Triamcinolone; Methylprednisolone; Shoulder pain
MeSH Terms: conditions — Shoulder Pain | interventions — Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Methylprednisolone, 20 mg (Active Comparator): Methylprednisolone, 20 mg, will be injected
  Interventions: Drug: Methylprednisolone, 40 mg
- Methylprednisolone, 40 mg (Active Comparator): Methylprednisolone, 40 mg, will be injected
  Interventions: Drug: Methylprednisolone, 20 mg
- Triamcinolone, 20 mg (Active Comparator): Triamcinolone, 20 mg, will be injected
  Interventions: Drug: Triamcinolone, 40 mg
- Triamcinolone, 40 mg (Active Comparator): Triamcinolone, 40 mg, will be injected
  Interventions: Drug: Triamcinolone, 20 mg

INTERVENTIONS:
Drug: Methylprednisolone, 20 mg — Compared with intrabursal triamcinolone
  Other Names: Depo-Medrol or Solu-Medrol
  Arms: Methylprednisolone, 40 mg
Drug: Methylprednisolone, 40 mg — Compared with intrabursal triamcinolone
  Other Names: Depo-Medrol or Solu-Medrol
  Arms: Methylprednisolone, 20 mg
Drug: Triamcinolone, 20 mg — Compared with methylprednisolone
  Other Names: Kenalog
  Arms: Triamcinolone, 40 mg
Drug: Triamcinolone, 40 mg — Compared with methylprednisolone
  Other Names: Kenalog
  Arms: Triamcinolone, 20 mg

SUMMARY:
It is currently unknown whether or not the improvement in pain and function related to a "steroid shot" for shoulder pain due to subacromial bursitis is important. This study seeks to determine whether 20 mg or 40 mg of either triamcinolone or methylprednisolone significantly affect improvement in shoulder pain 6 weeks after injection.

DETAILED DESCRIPTION:
Background: Subacromial bursitis is a common site for patients to report shoulder pain. In some patients it is refractory to conservative therapies such as physical therapy, acetaminophen, or NSAIDs. Subacromial injection of a corticosteroid can be used to improve shoulder pain in subacromial bursitis, however, there are few well done clinical trials guiding which type of corticosteroid and the dose that would be maximally effective and with the least amount of side effects.

Methods: Our hypothesis is that both Methylprednisolone and Triamcinolone are equipotent but that 20 mg provides less relief that 40 mg injected. Subjects will be enrolled in this trial which lasts 6 weeks. Subjects will be randomized to 40 mg of methylprednisolone, 20 mg of methylprednisolone, 40 mg of triamcinolone, or 20 mg of triamcinolone. No placebo will be used as prior studies suggest that placebo with lidocaine is inferior to corticosteroid injection.

Outcomes: Primary outcome with be the improvement in a functional measure of the shoulder, the QuickDASH ®, at 6 weeks. Secondary outcomes will be improvement in reported pain (visual analogue scale) at 6 weeks and adverse events at all time points. Data will be collected in person at the time of injection and then by phone at day 3, day 21 (3 weeks), and day 42 (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History and physical examination consistent with shoulder pain and subacromial bursitis
* At least 2 weeks of shoulder pain and subacromial bursitis

Exclusion Criteria:

* Known allergies to Lidocaine, Marcaine, Methylprednisolone, and/or Triamcinolone
* History or examination suspicious for a humeral head fracture
* History or examination consistent with adhesive capsulitis (normal X-Ray of the shoulder but with less than 100 degrees of active or passive elevation of the arm, when raising the arm above the head to a maximum with passive external rotation being 50 degrees less than the unaffected side
* History or examination consistent with acute synovitis of the glenohumeral or acromioclavicular joint
* Any shoulder surgery involving the affected arm within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Carroll, MD, Principal Investigator — Keesler Medical Center
Locations (1):
- Keesler Medical Center, Keesler Air Force Base, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
No plan to release IPD to other researchers

REFERENCES:
- [Derived] Carroll MB, Motley SA, Smith B, Ramsey BC, Baggett AS. Comparing Corticosteroid Preparation and Dose in the Improvement of Shoulder Function and Pain: A Randomized, Single-Blind Pilot Study. Am J Phys Med Rehabil. 2018 Jun;97(6):450-455. doi: 10.1097/PHM.0000000000000758. PMID 28609319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for this study were recruited from the internal medicine (IM) clinic or IM subspecialties clinic from our academic community hospital between September 2014 and December 2015. Subjects had to satisfy the inclusion criteria and have none of the exclusion criteria.
Pre-assignment Details: There was no wash out, run-in, or transitions in this trial.
Groups:
- Methylprednisolone, 20 mg: Methylprednisolone, 20 mg, will be injected
  Methylprednisolone, 40 mg: Compared with intrabursal triamcinolone
  Triamcinolone, 20 mg: Compared with methylprednisolone
  Triamcinolone, 40 mg: Compared with methylprednisolone
- Methylprednisolone, 40 mg: Methylprednisolone, 40 mg, will be injected
  Methylprednisolone, 20 mg: Compared with intrabursal triamcinolone
  Triamcinolone, 20 mg: Compared with methylprednisolone
  Triamcinolone, 40 mg: Compared with methylprednisolone
- Triamcinolone, 20 mg: Triamcinolone, 20 mg, will be injected
  Methylprednisolone, 20 mg: Compared with intrabursal triamcinolone
  Methylprednisolone, 40 mg: Compared with intrabursal triamcinolone
  Triamcinolone, 40 mg: Compared with methylprednisolone
- Triamcinolone, 40 mg: Triamcinolone, 40 mg, will be injected
  Methylprednisolone, 20 mg: Compared with intrabursal triamcinolone
  Methylprednisolone, 40 mg: Compared with intrabursal triamcinolone
  Triamcinolone, 20 mg: Compared with methylprednisolone
Period: Overall Study
Arm/Group | Methylprednisolone, 20 mg | Methylprednisolone, 40 mg | Triamcinolone, 20 mg | Triamcinolone, 40 mg
Started | 15 | 15 | 15 | 16
Completed | 15 | 15 | 15 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fifteen subjects were enrolled in each arm except for the TAC40 arm which had 16. The average age of the cohort was 67.1 ± 10.8 years old.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone, 20 mg | Methylprednisolone, 40 mg | Triamcinolone, 20 mg | Triamcinolone, 40 mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 7 | 8 | 31
  >=65 years | 7 | 7 | 8 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (10.9) | 69.3 (10.0) | 66.9 (12.3) | 69.0 (9.5) | 67.1 (10.8)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 6 | 6 | 7 | 29
  Male | 5 | 9 | 9 | 9 | 32
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 16 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Shoulder Function, as Measured by the QuickDASH ®
Description: The primary outcome of this study will be to compare the dose and type of intrabursal corticosteroid received to improvements in a functional measure of the shoulder, the QuickDASH. The QuickDASH is a validated questionnaire of shoulder function consisting of 11 questions with a score from 100 (maximal dysfunction) to 0 (no dysfunction). It is expected that improvements will lead to at least a 10 point improvement (minimal clinically important difference)
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methylprednisolone, 20 mg | Methylprednisolone, 40 mg | Triamcinolone, 20 mg | Triamcinolone, 40 mg
Number analyzed (Participants) | 15 | 15 | 15 | 16
units on a scale | 19.2 [7.1 to 31.4] | 21.3 [11.3 to 31.4] | 19.1 [11.8 to 26.4] | 24.7 [16.4 to 33.1]

2. Secondary Outcome: Change in Subject Reported Shoulder Pain as Measured by the Visual Analogue Scale
Description: Change in shoulder pain reported by the subject after injection at 6 weeks. The subject will report shoulder pain on a scale from 0 (no pain) to 10 (maximal pain) after injection. A 2 point change is expected.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methylprednisolone, 20 mg | Methylprednisolone, 40 mg | Triamcinolone, 20 mg | Triamcinolone, 40 mg
Number analyzed (Participants) | 15 | 15 | 15 | 16
units on a scale | 1.0 [0.1 to 1.9] | 1.8 [0.1 to 3.5] | 1.9 [0.6 to 3.2] | 1.8 [0.4 to 3.2]

3. Other Pre Specified Outcome: Safety
Description: Safety of either methylprednisolone or triamcinolone, either related to the medication received or the dose received.
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data regarding adverse events were collected for the 6 weeks that subjects were followed in this trial, with subjects queried about adverse events at the time of injection, 3 days after injection, 3 weeks, and 6 weeks after injection.
Arm/Group | Methylprednisolone, 20 mg | Methylprednisolone, 40 mg | Triamcinolone, 20 mg | Triamcinolone, 40 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 0/15 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylprednisolone, 20 mg (N=15) | Methylprednisolone, 40 mg (N=15) | Triamcinolone, 20 mg (N=15) | Triamcinolone, 40 mg (N=16)
Elevated blood glucose (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Increase in blood glucose as measured by participant which would be considered by the participant as beyond their normal range

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes